CLINICAL TRIAL: NCT07024641
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of GIGA-2339 Administered as a Single Ascending Dose and Multiple Ascending Doses in Participants With Chronic Hepatitis B Virus Infection
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of GIGA-2339 in Participants With Chronic Hepatitis B Virus Infection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GigaGen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GC2301
Record Dates: First submitted 2025-04-30; First posted 2025-06-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hepatitis B Virus Infection
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Single Ascending Dose (SAD) (Experimental): Participants will receive a single IV infusion of either GIGA-2339 or placebo in ascending doses on Day 1.
  Interventions: Drug: GIGA-2339; Drug: Placebo
- Part 2: Multiple Ascending Dose (MAD) (Experimental): Participants will receive multiple IV infusions of either GIGA-2339 or placebo, once every 4 weeks, at a dose determined in Part 1.
  Interventions: Drug: GIGA-2339; Drug: Placebo

INTERVENTIONS:
Drug: GIGA-2339 — Administered by intravenous infusion
Drug: Placebo — Administered by intravenous infusion

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of single and multiple intravenous (IV) doses of GIGA-2339 in participants with chronic Hepatitis B Virus (HBV) infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Hepatitis B envelope antigen (HBeAg) negative chronic HBV infection for ≥ 6 months, defined as presence of Hepatitis B surface antigen (HBsAg) in serum for ≥ 6 months.
* Serum HBsAg concentration between ≥ 100 international units per milliliter (IU/mL) and 2000 IU/mL at screening.
* Currently on stable dose of nucleot(s)ide analogues (NAs) (≥ 6 months) and expected to continue while participating in the study, or are not received NAs.
* Have serum HBV deoxyribonucleic acid (DNA) concentration ≤ 50 IU/mL at screening (for those who are on NAs); or have serum HBV DNA concentration ≤ 2000 IU/mL at screening (for those who are NOT on NAs).
* Male participants must refrain from donating spermatozoa and agree to use highly effective contraception.
* Female participants must not be pregnant, or breastfeeding; either should not be a woman of childbearing potential (WOCBP) or if WOCBP should use highly effective contraceptive methods.

Key Exclusion Criteria:

* Positive for co-infection with hepatitis C virus (HCV), human immunodeficiency virus (HIV), and/or hepatitis D virus (HDV) at screening.
* Participants that weigh less than 50 kilograms (kg) and/or have a body mass index (BMI) less than 18.5.
* History of documented liver cirrhosis at screening. Patients under liver cirrhosis evaluation at screening will not be eligible until cirrhosis is ruled out.
* Liver stiffness > 8 kilopascal (kPa) at screening.
* History of chronic liver disease from another cause, immune complex disease, or autoimmune diseases that in the opinion of the investigator would preclude participation.
* Family history of hepatocellular carcinoma (HCC).
* Alpha fetoprotein > 20 nanograms per milliliter (ng/mL).
* Presence of a liver imaging reporting and data system (LI-RADS) 4 or 5 liver lesion on imaging 12 months prior to Screening OR, LI-RADS-US findings of US-3 grade on imaging 12 months prior to Screening, OR LIRADS-US grade 3 done prior to the D1 infusion visit, if prior LI-RADS or LI-RADS-US results are not available at Screening.
* History of hematopoietic stem cell transplant or solid organ transplant.
* Receipt of anti-HBV monoclonal antibody (mAb)/pAb therapy of any kind in the past (including hepatitis B immunoglobulin [HBIG]).
* History of cardiovascular disease (e.g., coronary artery disease, cardiomyopathy, congestive heart failure, family history of congenital long QT syndrome). Stable hypertension is allowed.
* Malignancy diagnosed and/or treated within 5 years prior to Screening, and/or with ongoing treatment for malignancy, with the exception of localized non-metastatic basal cell or squamous cell carcinoma of the skin or in-situ carcinoma of the cervix excised with curative intent.
* Participants requiring anti-coagulation therapies (for example warfarin, Factor Xa inhibitors, or anti-platelet agents like clopidogrel).
* Male participants with a corrected QT interval using Fridericia's formula (QTcF) > 450 milliseconds (msec) and female participants with QTcF > 470 msec on ECG recorded at screening. if the participant has evidence of an intraventricular conduction delay, defined as QRS interval greater than 110 msec, a QTcF is > 500 msec for both males and females will be excluded.
* Known hypersensitivity to any GIGA-2339 excipients or any confirmed significant allergic reactions (urticaria or anaphylaxis) against any drug, or multiple drug allergies (nonactive hay fever is acceptable), or a history of drug or other allergy that, in the opinion of the Investigator, contraindicates participation.
* Received or will receive live-attenuated virus vaccinations such as measles, mumps, rubella or varicella within 4 weeks before and up to three months after administration of investigational product (IP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
SAD and MAD: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | SAD: Up to Day 105; MAD: Up to Day 245

SECONDARY OUTCOMES:
SAD and MAD: Maximum Serum Concentration (Cmax) of GIGA-2339 | SAD: Pre-dose and at multiple timepoints post-dose up to Day 105; MAD: Pre-dose and at multiple timepoints post-dose up to Day 245
SAD and MAD: Area Under the Concentration Time Curve (AUC) from 0 to the Last Quantifiable Concentration (AUC0-t) of GIGA-2339 | SAD: Pre-dose and at multiple timepoints post-dose up to Day 105; MAD: Pre-dose and at multiple timepoints post-dose up to Day 245
SAD: AUC From 0 to Infinity (AUC0-∞) of GIGA-2339 | Pre-dose and at multiple timepoints post-dose up to Day 105
SAD: Dose Normalized Maximum Serum Concentration (DN_Cmax). of GIGA-2339 | Pre-dose and at multiple timepoints post-dose up to Day 105
SAD: Dose Normalized AUC From 0 to the Last Quantifiable Concentration (DN_AUC0-t) of GIGA-2339 | Pre-dose and at multiple timepoints post-dose up to Day 105
SAD: Dose Normalized AUC From 0 to Infinity (DN_AUC0-∞) of GIGA-2339 | Pre-dose and at multiple timepoints post-dose up to Day 105
SAD and MAD: Time to Obtain Maximum Concentration (Tmax) of GIGA-2339 | SAD: Pre-dose and at multiple timepoints post-dose up to Day 105; MAD: Pre-dose and at multiple timepoints post-dose up to Day 245
SAD and MAD: Terminal Half-Life (t1/2) of GIGA-2339 | SAD: Pre-dose and at multiple timepoints post-dose up to Day 105; MAD: Pre-dose and at multiple timepoints post-dose up to Day 245
SAD and MAD: Volume of Distribution (Vz) of GIGA-2339 | SAD: Pre-dose and at multiple timepoints post-dose up to Day 105; MAD: Pre-dose and at multiple timepoints post-dose up to Day 245
SAD and MAD: Systemic Clearance (CL) of GIGA-2339 | SAD: Pre-dose and at multiple timepoints post-dose up to Day 105; MAD: Pre-dose and at multiple timepoints post-dose up to Day 245
MAD: Serum Concentration at the End of the Dosing Interval (Ctrough) of GIGA-2339 | Pre-dose and at multiple timepoints post-dose up to Day 245
MAD: AUC Versus Time Curve During the Dosing Interval (AUC0-tau) of GIGA-2339 | Pre-dose and at multiple timepoints post-dose up to Day 245
MAD: Accumulation Ratio Cmax (ARCmax) of GIGA-2339 | Pre-dose and at multiple timepoints post-dose up to Day 245
MAD: Accumulation Ratio AUC (ARAUCs) of GIGA-2339 | Pre-dose and at multiple timepoints post-dose up to Day 245

CONTACTS AND LOCATIONS:
Locations (14):
- United States (12):
  - Grifols Investigative site, Chandler, Arizona
  - Grifols Investigative site, Huntington Beach, California
  - Grifols Investigative site, Lake Forest, California
  - Grifols Investigative site, Long Beach, California
  - Grifols Investigative site, Oakland, California
  - Grifols Investigative Site, Peachtree Corners, Georgia
  - Grifols Investigative Site, Iowa City, Iowa
  - Grifols Investigative Site, Lenexa, Kansas
  - Grifols Investigative site, Baltimore, Maryland
  - Grifols Investigative site, San Antonio, Texas
  - Grifols Investigative site, Webster, Texas
  - Grifols Investigative site, Richmond, Virginia
- Australia (2):
  - Grifols Investigate Site, Concord, New South Wales
  - Grifols Investigative site, Fortitude Valley, Queensland

IPD SHARING:
Plan to Share IPD: Undecided